CLINICAL TRIAL: NCT05017519
Title: Epidemiology and Transmission of Streptococcus Pneumoniae and Respiratory Syncytial Virus in Children and Elderly: a Household-based Prospective Cohort Study
Brief Title: Epidemiology and Household Transmission of Streptococcus Pneumoniae and Respiratory Syncytial Virus
Status: Not yet recruiting | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Hsin Chi, Dr., Mackay Memorial Hospital
Other Study IDs: MSD MISP 60284
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Streptococcus Pneumoniae Infection; Respiratory Syncytial Virus Infections
Keywords: Streptococcus Pneumoniae; Respiratory Syncytial Virus; household-based
MeSH Terms: conditions — Pneumococcal Infections; Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Nasopharyngeal or throat swab and urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nuclear family type: The husband and wife with baby (aged less than 5 months) and with or without children (2-5)
- Extended family type (three-generation family): The husband and wife with baby (aged less than 5 months), children (2-5), and grandparents aged > 65 years old

SUMMARY:
This household-based prospective cohort study aims to stablish the household transmission of Respiratory syncytial virus and S. pneumoniae especially in the elderly and infants/children as well as inter-relationship between S. pneumoniae and Respiratory syncytial virus.

DETAILED DESCRIPTION:
A household-based prospective cohort study will be conducted from 2021 to 2025 in northern Taiwan. We will invite 240 households, having a baby who is discharged from MacKay children's Hospital. The households will be classified into nuclear family type and extended family type. The "Nuclear family type" is defined as husband and wife with baby (aged less than 5 months) and with or without children (2-5) and the "Extended family type" (three-generation family) is defined as husband and wife with baby (aged less than 5 months), children (2-5), and grandparents aged > 65 years old. We will initially complete an enrollment form to collect baseline data, including patient demographics, prior medical history, season when discharge, neonatal course and households. A LINE-based management will be done weekly by study team to see if there are any respiratory symptoms in household. In addition to the monthly physician weekly LINE response, the research nurse will contact the parents or legal guardians by telephone monthly for the 24 months to obtain data on changes in baseline information, and specific facts regarding possible respiratory infections after the last contact. If the households present with respiratory symptoms, the visit will be arranged as early as possible. When they presenting to the emergency department, outpatient clinic, or inpatient ward, the urine will be collected for the serotype-specific urinary antigen detection (SSUAD) assays and the nasopharyngeal or throat swab for polymerase chain reaction will be performed to study serotype of S. pneumoniae and Respiratory syncytial virus subgroup. If the subjects who have clinical syndromes suggestive of pneumonia or bronchopneumonia, they will be asked to participate in the further study along with their household family members. Nasopharyngeal aspiration, urine, blood, and induced sputum will be collected for cultures, polymerase chain reaction and serological test. Clinical manifestations, disease course, and outcomes will be recorded. Family members in the same household will asked to undergo screening with a nasopharyngeal or throat swab and urine sample. We will trace back 2-week contact history of children in nuclear family who get Respiratory syncytial virus or pneumococcal infections, especially focus on other family members. The data will be further analyzed to evaluate the influence of short period and long period contact.

ELIGIBILITY:
Inclusion Criteria:

* Indicator case: Babies under 5 months of age were born in Mackay Children's Hospital and had no acute respiratory infection-like symptoms that required medical intervention when they agreed to participate in the trial.
* Family members: family members living with the Indicator case, including 2-5 years old siblings, parents and grandparents over 65 years old.
* Willing to sign the informed consent form and agree to join the official LINE account to receive research tracking.

Exclusion Criteria:

* Babies older than 5 months
* Co-morbid medical conditions of the baby such as chronic lung disease, cyanotic congenital heart disease, neuromuscular disease and a primary immunodeficiency.
* Family members who do not live with the Indicator case
* Family with grandparents younger than 65 years old
* Someone living with family members refuses to participate in the research.
* Unwilling to sign informed consent form or refuse to join the official LINE account to receive tracking.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A household-based prospective cohort study will invite 240 households, having a baby who is discharged from MacKay children's Hospital. The households will be classified into nuclear family type and extended family type. The "Nuclear family type" is defined as husband and wife with baby (aged less than 5 months) and with or without children (2-5) and the "Extended family type" (three-generation family) is defined as husband and wife with baby (aged less than 5 months), children (2-5), and grandparents aged > 65 years old.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Household transmission of Streptococcus pneumoniae and Respiratory syncytial virus | 2 years
  The primary endpoint is the Streptococcus pneumoniae and Respiratory syncytial virus isolation rates in children and their household contacts of different family type.
The serotype of Streptococcus pneumoniae and Respiratory syncytial virus in post-Prevenar 13 era | 2 years
  The secondary endpoint is the serotype of Streptococcus pneumoniae and Respiratory syncytial virus in post-Prevenar 13 era.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin Chi, Doctor, Principal Investigator — Mackay Children's Hospital in Taiwan

IPD SHARING:
Plan to Share IPD: No
We will record and analyze the individual participant data by our study team only.

REFERENCES:
- [Result] Huang YC, Lin CF, Ting PJ, Tang TH, Huang FL, Chao HJ, Wang CL, Chen PY. Respiratory pathogens - Some altered antibiotic susceptibility after implementation of pneumococcus vaccine and antibiotic control strategies. J Microbiol Immunol Infect. 2020 Oct;53(5):682-689. doi: 10.1016/j.jmii.2019.08.015. Epub 2019 Oct 18. PMID 31859164
- [Result] Lu CY, Chiang CS, Chiu CH, Wang ET, Chen YY, Yao SM, Chang LY, Huang LM, Lin TY, Chou JH. Successful Control of Streptococcus pneumoniae 19A Replacement With a Catch-up Primary Vaccination Program in Taiwan. Clin Infect Dis. 2019 Oct 15;69(9):1581-1587. doi: 10.1093/cid/ciy1127. PMID 30923808
- [Result] Feikin DR, Kagucia EW, Loo JD, Link-Gelles R, Puhan MA, Cherian T, Levine OS, Whitney CG, O'Brien KL, Moore MR; Serotype Replacement Study Group. Serotype-specific changes in invasive pneumococcal disease after pneumococcal conjugate vaccine introduction: a pooled analysis of multiple surveillance sites. PLoS Med. 2013;10(9):e1001517. doi: 10.1371/journal.pmed.1001517. Epub 2013 Sep 24. PMID 24086113
- [Result] Chi HC, Hsieh YC, Tsai MH, Lee CH, Kuo KC, Huang CT, Huang YC. Impact of pneumococcal conjugate vaccine in children on the serotypic epidemiology of adult invasive pneumococcal diseases in Taiwan. J Microbiol Immunol Infect. 2018 Jun;51(3):332-336. doi: 10.1016/j.jmii.2016.08.009. Epub 2016 Dec 18. PMID 28082066
- [Result] Ladhani SN, Collins S, Djennad A, Sheppard CL, Borrow R, Fry NK, Andrews NJ, Miller E, Ramsay ME. Rapid increase in non-vaccine serotypes causing invasive pneumococcal disease in England and Wales, 2000-17: a prospective national observational cohort study. Lancet Infect Dis. 2018 Apr;18(4):441-451. doi: 10.1016/S1473-3099(18)30052-5. Epub 2018 Jan 26. PMID 29395999
- [Result] Hall CB, Weinberg GA, Iwane MK, Blumkin AK, Edwards KM, Staat MA, Auinger P, Griffin MR, Poehling KA, Erdman D, Grijalva CG, Zhu Y, Szilagyi P. The burden of respiratory syncytial virus infection in young children. N Engl J Med. 2009 Feb 5;360(6):588-98. doi: 10.1056/NEJMoa0804877. PMID 19196675
- [Result] Obando-Pacheco P, Justicia-Grande AJ, Rivero-Calle I, Rodriguez-Tenreiro C, Sly P, Ramilo O, Mejias A, Baraldi E, Papadopoulos NG, Nair H, Nunes MC, Kragten-Tabatabaie L, Heikkinen T, Greenough A, Stein RT, Manzoni P, Bont L, Martinon-Torres F. Respiratory Syncytial Virus Seasonality: A Global Overview. J Infect Dis. 2018 Apr 11;217(9):1356-1364. doi: 10.1093/infdis/jiy056. PMID 29390105
- [Result] Lin CY, Hwang D, Chiu NC, Weng LC, Liu HF, Mu JJ, Liu CP, Chi H. Increased Detection of Viruses in Children with Respiratory Tract Infection Using PCR. Int J Environ Res Public Health. 2020 Jan 15;17(2):564. doi: 10.3390/ijerph17020564. PMID 31952364
- [Result] Pneumonia Etiology Research for Child Health (PERCH) Study Group. Causes of severe pneumonia requiring hospital admission in children without HIV infection from Africa and Asia: the PERCH multi-country case-control study. Lancet. 2019 Aug 31;394(10200):757-779. doi: 10.1016/S0140-6736(19)30721-4. Epub 2019 Jun 27. PMID 31257127
- [Result] Wolf DG, Greenberg D, Shemer-Avni Y, Givon-Lavi N, Bar-Ziv J, Dagan R. Association of human metapneumovirus with radiologically diagnosed community-acquired alveolar pneumonia in young children. J Pediatr. 2010 Jan;156(1):115-20. doi: 10.1016/j.jpeds.2009.07.014. PMID 19782998
- [Result] Jain S, Williams DJ, Arnold SR, Ampofo K, Bramley AM, Reed C, Stockmann C, Anderson EJ, Grijalva CG, Self WH, Zhu Y, Patel A, Hymas W, Chappell JD, Kaufman RA, Kan JH, Dansie D, Lenny N, Hillyard DR, Haynes LM, Levine M, Lindstrom S, Winchell JM, Katz JM, Erdman D, Schneider E, Hicks LA, Wunderink RG, Edwards KM, Pavia AT, McCullers JA, Finelli L; CDC EPIC Study Team. Community-acquired pneumonia requiring hospitalization among U.S. children. N Engl J Med. 2015 Feb 26;372(9):835-45. doi: 10.1056/NEJMoa1405870. PMID 25714161
- [Result] Chiu NC, Lin HY, Hsu CH, Huang FY, Lee KS, Chi H. Epidemiological and microbiological characteristics of culture-proven acute otitis media in Taiwanese children. J Formos Med Assoc. 2012 Oct;111(10):536-41. doi: 10.1016/j.jfma.2011.07.015. Epub 2012 Mar 13. PMID 23089688
- [Result] Kung YH, Chiu NC, Lee KS, Chang L, Huang DT, Huang FY, Hsieh YC, Huang LM, Chi H. Bacterial etiology of acute otitis media in the era prior to universal pneumococcal vaccination in Taiwanese children. J Microbiol Immunol Infect. 2014 Jun;47(3):239-44. doi: 10.1016/j.jmii.2013.08.016. Epub 2013 Sep 27. PMID 24080520
- [Result] Patel JA, Nguyen DT, Revai K, Chonmaitree T. Role of respiratory syncytial virus in acute otitis media: implications for vaccine development. Vaccine. 2007 Feb 19;25(9):1683-9. doi: 10.1016/j.vaccine.2006.10.045. Epub 2006 Nov 9. PMID 17156899
- [Result] de Steenhuijsen Piters WA, Heinonen S, Hasrat R, Bunsow E, Smith B, Suarez-Arrabal MC, Chaussabel D, Cohen DM, Sanders EA, Ramilo O, Bogaert D, Mejias A. Nasopharyngeal Microbiota, Host Transcriptome, and Disease Severity in Children with Respiratory Syncytial Virus Infection. Am J Respir Crit Care Med. 2016 Nov 1;194(9):1104-1115. doi: 10.1164/rccm.201602-0220OC. PMID 27135599
- [Result] Tsolia MN, Psarras S, Bossios A, Audi H, Paldanius M, Gourgiotis D, Kallergi K, Kafetzis DA, Constantopoulos A, Papadopoulos NG. Etiology of community-acquired pneumonia in hospitalized school-age children: evidence for high prevalence of viral infections. Clin Infect Dis. 2004 Sep 1;39(5):681-6. doi: 10.1086/422996. Epub 2004 Aug 13. PMID 15356783
- [Result] Ampofo K, Bender J, Sheng X, Korgenski K, Daly J, Pavia AT, Byington CL. Seasonal invasive pneumococcal disease in children: role of preceding respiratory viral infection. Pediatrics. 2008 Aug;122(2):229-37. doi: 10.1542/peds.2007-3192. PMID 18676537
- [Result] Brealey JC, Chappell KJ, Galbraith S, Fantino E, Gaydon J, Tozer S, Young PR, Holt PG, Sly PD. Streptococcus pneumoniae colonization of the nasopharynx is associated with increased severity during respiratory syncytial virus infection in young children. Respirology. 2018 Feb;23(2):220-227. doi: 10.1111/resp.13179. Epub 2017 Sep 15. PMID 28913912
- [Result] Nguyen DT, Louwen R, Elberse K, van Amerongen G, Yuksel S, Luijendijk A, Osterhaus AD, Duprex WP, de Swart RL. Streptococcus pneumoniae Enhances Human Respiratory Syncytial Virus Infection In Vitro and In Vivo. PLoS One. 2015 May 13;10(5):e0127098. doi: 10.1371/journal.pone.0127098. eCollection 2015. PMID 25970287
- [Result] Greenberg D, Givon-Lavi N, Faingelernt Y, Ben-Shimol S, Avni YS, Bar-Ziv J, Dagan R. Nasopharyngeal Pneumococcal Carriage During Childhood Community-Acquired Alveolar Pneumonia: Relationship Between Specific Serotypes and Coinfecting Viruses. J Infect Dis. 2017 Apr 1;215(7):1111-1116. doi: 10.1093/infdis/jiw613. PMID 28011920
- [Result] Althouse BM, Hammitt LL, Grant L, Wagner BG, Reid R, Larzelere-Hinton F, Weatherholtz R, Klugman KP, Rodgers GL, O'Brien KL, Hu H. Identifying transmission routes of Streptococcus pneumoniae and sources of acquisitions in high transmission communities. Epidemiol Infect. 2017 Oct;145(13):2750-2758. doi: 10.1017/S095026881700125X. Epub 2017 Aug 29. PMID 28847317
- [Result] Tramuto F, Amodio E, Calamusa G, Restivo V, Costantino C, Vitale F; The BINOCOLO Group. Pneumococcal Colonization in the Familial Context and Implications for Anti-Pneumococcal Immunization in Adults: Results from the BINOCOLO Project in Sicily. Int J Mol Sci. 2017 Jan 6;18(1):105. doi: 10.3390/ijms18010105. PMID 28067813
- [Result] Walsh EE, Falsey AR. Respiratory syncytial virus infection in adult populations. Infect Disord Drug Targets. 2012 Apr;12(2):98-102. doi: 10.2174/187152612800100116. PMID 22335500
- [Result] Agoti CN, Munywoki PK, Phan MVT, Otieno JR, Kamau E, Bett A, Kombe I, Githinji G, Medley GF, Cane PA, Kellam P, Cotten M, Nokes DJ. Transmission patterns and evolution of respiratory syncytial virus in a community outbreak identified by genomic analysis. Virus Evol. 2017 Mar 11;3(1):vex006. doi: 10.1093/ve/vex006. eCollection 2017 Jan. PMID 28458916
- [Result] Crowcroft NS, Zambon M, Harrison TG, Mok Q, Heath P, Miller E. Respiratory syncytial virus infection in infants admitted to paediatric intensive care units in London, and in their families. Eur J Pediatr. 2008 Apr;167(4):395-9. doi: 10.1007/s00431-007-0509-9. Epub 2007 May 31. PMID 17541638
- [Result] Otomaru H, Kamigaki T, Tamaki R, Okamoto M, Alday PP, Tan AG, Manalo JI, Segubre-Mercado E, Inobaya MT, Tallo V, Lupisan S, Oshitani H. Transmission of Respiratory Syncytial Virus Among Children Under 5 Years in Households of Rural Communities, the Philippines. Open Forum Infect Dis. 2019 Mar 11;6(3):ofz045. doi: 10.1093/ofid/ofz045. eCollection 2019 Mar. PMID 30882012
- [Result] Munywoki PK, Koech DC, Agoti CN, Lewa C, Cane PA, Medley GF, Nokes DJ. The source of respiratory syncytial virus infection in infants: a household cohort study in rural Kenya. J Infect Dis. 2014 Jun 1;209(11):1685-92. doi: 10.1093/infdis/jit828. Epub 2013 Dec 23. PMID 24367040
- [Result] Kim L, Rha B, Abramson JS, Anderson LJ, Byington CL, Chen GL, DeVincenzo J, Edwards KM, Englund JA, Falsey AR, Griffin MR, Karron RA, Martin KG, Meissner HC, Munoz FM, Pavia AT, Piedra PA, Schaffner W, Simoes EAF, Singleton R, Talbot HK, Walsh EE, Zucker JR, Gerber SI. Identifying Gaps in Respiratory Syncytial Virus Disease Epidemiology in the United States Prior to the Introduction of Vaccines. Clin Infect Dis. 2017 Sep 15;65(6):1020-1025. doi: 10.1093/cid/cix432. PMID 28903503
- [Result] Midgley CM, Haynes AK, Baumgardner JL, Chommanard C, Demas SW, Prill MM, Abedi GR, Curns AT, Watson JT, Gerber SI. Determining the Seasonality of Respiratory Syncytial Virus in the United States: The Impact of Increased Molecular Testing. J Infect Dis. 2017 Aug 1;216(3):345-355. doi: 10.1093/infdis/jix275. PMID 28859428
- [Result] Smith CM, Sandrini S, Datta S, Freestone P, Shafeeq S, Radhakrishnan P, Williams G, Glenn SM, Kuipers OP, Hirst RA, Easton AJ, Andrew PW, O'Callaghan C. Respiratory syncytial virus increases the virulence of Streptococcus pneumoniae by binding to penicillin binding protein 1a. A new paradigm in respiratory infection. Am J Respir Crit Care Med. 2014 Jul 15;190(2):196-207. doi: 10.1164/rccm.201311-2110OC. PMID 24941423
- [Result] Yan T, Tang X, Sun L, Tian R, Li Z, Liu G. Co infection of respiratory syncytial viruses (RSV) and streptococcus pneumonia modulates pathogenesis and dependent of serotype and phase variant. Microb Pathog. 2020 Jul;144:104126. doi: 10.1016/j.micpath.2020.104126. Epub 2020 Mar 12. PMID 32173494 (Retraction: PMID 35400546 Microb Pathog. 2022 Apr;165:105486)
- [Result] Chi H, Liu HF, Weng LC, Wang NY, Chiu NC, Lai MJ, Lin YC, Chiu YY, Hsieh WS, Huang LM. Molecular epidemiology and phylodynamics of the human respiratory syncytial virus fusion protein in northern Taiwan. PLoS One. 2013 May 29;8(5):e64012. doi: 10.1371/journal.pone.0064012. Print 2013. PMID 23734183
- [Result] Pai R, Gertz RE, Beall B. Sequential multiplex PCR approach for determining capsular serotypes of Streptococcus pneumoniae isolates. J Clin Microbiol. 2006 Jan;44(1):124-31. doi: 10.1128/JCM.44.1.124-131.2006. PMID 16390959
- [Result] Leung MH, Bryson K, Freystatter K, Pichon B, Edwards G, Charalambous BM, Gillespie SH. Sequetyping: serotyping Streptococcus pneumoniae by a single PCR sequencing strategy. J Clin Microbiol. 2012 Jul;50(7):2419-27. doi: 10.1128/JCM.06384-11. Epub 2012 May 2. PMID 22553238
- [Result] Melegaro A, Gay NJ, Medley GF. Estimating the transmission parameters of pneumococcal carriage in households. Epidemiol Infect. 2004 Jun;132(3):433-41. doi: 10.1017/s0950268804001980. PMID 15188713
- [Result] Menashe I, Rosenberg PS, Chen BE. PGA: power calculator for case-control genetic association analyses. BMC Genet. 2008 May 13;9:36. doi: 10.1186/1471-2156-9-36. PMID 18477402
- [Result] Erasto P, Hoti F, Auranen K. Modeling transmission of multitype infectious agents: application to carriage of Streptococcus pneumoniae. Stat Med. 2012 Jun 30;31(14):1450-63. doi: 10.1002/sim.4487. Epub 2012 Feb 21. PMID 22354452
- [Result] Chang LY, Tsao KC, Hsia SH, Shih SR, Huang CG, Chan WK, Hsu KH, Fang TY, Huang YC, Lin TY. Transmission and clinical features of enterovirus 71 infections in household contacts in Taiwan. JAMA. 2004 Jan 14;291(2):222-7. doi: 10.1001/jama.291.2.222. PMID 14722149
- [Result] Wang KS, Liu X, Ategbole M, Xie X, Liu Y, Xu C, Xie C, Sha Z. Generalized Linear Mixed Model Analysis of Urban-Rural Differences in Social and Behavioral Factors for Colorectal Cancer Screening. Asian Pac J Cancer Prev. 2017 Sep 27;18(9):2581-2589. doi: 10.22034/APJCP.2017.18.9.2581. PMID 28952708
- [Result] Glorioso TJ, Grunwald GK, Ho PM, Maddox TM. Reference effect measures for quantifying, comparing and visualizing variation from random and fixed effects in non-normal multilevel models, with applications to site variation in medical procedure use and outcomes. BMC Med Res Methodol. 2018 Jul 6;18(1):74. doi: 10.1186/s12874-018-0517-7. PMID 29980180

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT05017519/Prot_SAP_000.pdf